CLINICAL TRIAL: NCT06987630
Title: Effect of Continuous Integrated Pulmonary Index Monitoring on the Incidence of Hypoxemia in Elderly Patients With Painless Colonoscopy
Brief Title: Integrated Pulmonary Index Monitoring on the Incidence of Hypoxemia in Elderly Patients With Painless Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The First People's Hospital of Lianyungang (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: KY-20241226001-01
Record Dates: First submitted 2025-05-05; First posted 2025-05-23 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Hypoxia
Keywords: Elderly patients; Colonoscopy; Propofol
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- P group (Experimental): Nasal cannula oxygen inhalation, oxygen flow rate 3-4L/min, monitor the integrated pulmonary index and SpO2.
  Interventions: Device: monitor integrated pulmonary index（IPI） and take appropriate measures
- C group (No Intervention): Nasal cannula oxygen inhalation, oxygen flow rate 3-4L/min,monitor the SpO2,

INTERVENTIONS:
Device: monitor integrated pulmonary index（IPI） and take appropriate measures — When the IPI is ≤ 6, the patient's jaw is immediately lifted, the oxygen flow rate increases to 6L·min-1, and if the SpO2 continues to decrease by <90%, the anesthesia mask is pressurized and ventilated.
  Arms: P group

SUMMARY:
The purpose of this clinical trial is to integrated pulmonary index to see if there is an effect on the incidence of hypoxemia during painless colonoscopy in older patients.

Does composite pulmonary index monitoring reduce the incidence of hypoxemia? Is there a relationship between the value of the integrated pulmonary index and the patient's pulse oximetry? Continuous monitoring of the integrated pulmonary index in the experimental group was compared with the control group (no detection of the composite lung index) to see if continuous monitoring of the composite pulmonary index could reduce the incidence of hypoxemia in elderly patients.

Participants will:

Oxygen is provided through the nasal cannula, and respiratory parameters (end-tidal carbon dioxide partial pressure (PetCO2), pulse rate [PR], oxygen saturation (SpO2), and respiratory rate (RR) are obtained. The monitor calculates a integrated pulmonary index value (1-10) through mathematical operations.Different measures are taken according to different composite lung indexes, such as when the IPI is ≤6, the patient's jaw is immediately lifted, the oxygen flow rate increases to 6L·min-1, and if the SpO2 continues to decrease by <90%, the anesthesia mask is pressurized and ventilated.

Record their vital signs.

DETAILED DESCRIPTION:
This study is a single-center, double-blind, prospective, randomized controlled trial. In this experiment, all patients who met the inclusion criteria and did not meet any of the exclusion criteria were divided into SpO2 group (group C) and IPI group (group P) according to 1:1 by computer random number method. After entering the examination room, the two groups of patients signed the informed consent form and underwent vital sign monitoring. Anesthesia process: propofol 1~ 2mg/kg, Intraoperatively, vasoactive drugs such as norepinephrine or ephedrine are used as needed. Group C: SpO2 of the patient's right index finger was monitored with a fingertip oximeter. When the SpO2 decreases by 5% compared with the basic SpO2, the patient's jaw is immediately propped up, and the oxygen flow rate increases to 6L·min-1, and if the SpO2 continues to decrease by <90%, the anesthesia mask is pressurized and ventilated. Group P: Fingertip oximetry was used to monitor the SpO2 of the patient's right index finger, and the patient's PETCO2 was monitored with nasal cannula bypass, and when the IPI was ≤6, The patient's jaw is immediately lifted, the oxygen flow rate is increased to 6L·min-1, and if the SpO2 continues to decrease by <90%, the anesthesia mask is pressurized and ventilated. Vital signs (blood pressure, heart rate, pulse oximetry or IPI), medication (propofol or vasoactive), anesthesia time and adverse events were recorded in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were selected for non-intubated painless colonoscopy;
* Age≥ 65 years;
* American Society of Anesthesiologists (ASA) grade I~III;
* Conscious, no cognitive dysfunction and other mental illnesses;
* Voluntarily participate in this study and sign the informed consent form

Exclusion Criteria:

* Patients with severe circulatory system diseases, respiratory diseases, and central nervous system diseases;
* Patients with severe abnormal liver and kidney function;
* Those who are allergic to any of the drugs used in the study;
* Participated in other clinical studies within the last 3 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 153 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | Perioperative
  the number of patients experiencing low blood pressure

SECONDARY OUTCOMES:
Adverse reactions (dizziness, nausea, vomiting, etc.) | Perioperative
  The number of adverse reactions (dizziness, nausea, vomiting, etc.)

CONTACTS AND LOCATIONS:
Locations (1):
- The First People's Hospital of Lianyungang City, Lianyungang, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No